CLINICAL TRIAL: NCT04951583
Title: Phase II Trial of Fecal Microbial Transplantation in Patients With Advanced Non-Small Cell Lung Cancer and Melanoma Treated With Immune Checkpoint Inhibitors.
Brief Title: Fecal Microbial Transplantation Non-Small Cell Lung Cancer and Melanoma
Acronym: FMT-LUMINATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21.173
Record Dates: First submitted 2021-06-18; First posted 2021-07-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Advanced Melanoma
Keywords: FMT, ICI, Advanced NSCLC, advanced melanoma
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a multi-center single-arm, open-label Simon two-stage, phase II trial in patients with metastatic or unresectable non-small cell lung cancer (NSCLC) and melanoma treated with immune checkpoint inhibition.
  Patients will receive standard-of-care immune checkpoint inhibitor (ICI) therapy in combination with fecal microbial transplantation (FMT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immune checkpoint inhibitor (ICI) therapy in combination with fecal microbial transplantation (FMT). (Experimental): Metastatic or advanced NSCLC: Single-agent Pembrolizumab (2 mg/kg or 200 mg every 3 weeks) in combination with investigational FMT capsules as follows: Full FMT at least 7 days prior to first cycle of Pembrolizumab.
  Metastatic melanoma and uveal melanoma: Combination therapy of Ipilimumab plus Nivolumab (Ipilimumab 3 mg/kg every 3 weeks and Nivolumab 1 mg/kg every 3 weeks x 4 doses, followed by Nivolumab 3 mg/kg or 240mg every 2 weeks or 6 mg/kg or 480mg every 4 weeks) in combination with investigational FMT capsules as follows: full FMT at least 7 days prior to first treatment with Ipilimumab plus Nivolumab, followed by supportive FMT within 7 days of the second cycle with combination Ipilimumab plus Nivolumab, followed by supportive FMT within 7 days of the third cycle of Ipilimumab plus Nivolumab.
  Interventions: Combination Product: FMT + ICI

INTERVENTIONS:
Combination Product: FMT + ICI — This study will include 3 cohorts of patients: (1) Patients with advanced or unresectable NSCLC, (2) patients with advanced or unresectable melanoma, and (3) patients with unresectable or advanced uveal melanoma. Patients with NSCLC, melanoma, uveal melanoma and will be analyzed in three separate subgroups given their differing clinical outcomes.
  Each group will be treated with ICI as per their respective first line options, in combination with investigational FMT capsules.

SUMMARY:
The aim of this study is to assess the anti-tumor activity of FMT administered in combination with ICI therapy.

DETAILED DESCRIPTION:
Immune-checkpoint inhibitors (ICI) now represent the backbone therapy for patients with advanced or unresectable non-small cell lung cancer (NSCLC) and melanoma. With the use of anti-PD-1 (Pembrolizumab), overall survival (OS) is now 45% at two years for patients with metastatic NSCLC with a PD-L1 expression level above 50%. The OS for patients with metastatic melanoma is now 52% at five years with combination therapy of anti-CLTA-4 (Ipilimumab) and anti-PD-1 (Nivolumab).

However, only a minority of patients obtain durable responses and current biomarkers are unable to consistently and accurately predict response to ICI. Addressing these unmet needs, the gut microbiome has emerged as a potential biomarker of response to ICI. Modulating the gut microbiome to improve response to ICI is an active area of study. One way to modify the gut microbiome composition is through fecal microbial transplantation (FMT) and pre-clinical studies showed improved effectiveness of ICI when mice received FMT from lung cancer patients responding to ICI. Recently, 2 phase I clinical studies published in Science consolidated these findings, and demonstrated the safety of FMT in patients with melanoma treated with ICI.

Building on phase I studies showing that FMT is safe in patients with cancer receiving ICI, and compelling data demonstrating the potential of FMT to reverse ICI resistance, there is a strong rationale to further study the role of FMT in improving ICI efficacy in patients with melanoma and NSCLC treated with ICI in the first-line setting in a phase II study.

Our primary objective is to assess the impact of FMT on ICI response and survival. Other goals of this trial are to study the changes in the patient's gut microbiome composition and tumor microenvironment contexture following the combination treatment of ICI and FMT. Efficacy of FMT in terms of response rate and overall survival in patients with metastatic melanoma and uveal melanoma will be studies as part of an exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent;
2. Patients must be able to understand the infectious and non-infectious risks associated with FMT administration;
3. Must understand that data regarding the long-term safety risks of FMT administration are lacking;
4. Age 18 years or older;
5. Confirmed histological diagnosis of either: unresectable or metastatic melanoma, unresectable or metastatic uveal melanoma, or unresectable or metastatic non-small cell lung cancer (NSCLC);
6. Stage IV or unresectable disease;
7. No prior anti-PD1 treatment;
8. For patients with newly diagnosed metastatic melanoma who relapsed after adjuvant immunotherapy, patients can be included in this study if they relapsed >6 months after their last dose of immunotherapy given in the adjuvant setting;
9. For patients with NSCLC, tumor PD-L1 expression level 50%
10. Evaluable disease as per iRECIST;
11. ECOG performance status of 0-2;
12. Ability to ingest capsules;
13. Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (< 10 mg prednisone daily or equivalent permitted);
14. Negative pregnancy test for women of child-bearing potential; and
15. Highly effective contraception for both male and female subjects throughout the study and for at least 60 days after last treatment administration if the risk of conception exists

Exclusion Criteria:

1. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
2. Current or recent [in the last 90 days] exposure to high dose oral or IV corticosteroids

   a. Patients who require intermittent use of bronchodilators or local steroid injections are not excluded from the study.
3. Has a diagnosis of immunodeficiency (e.g. HIV, transplantation) or receiving systemic steroid therapy (>10mg prednisone daily or equivalent) or any other form of immunosuppressive therapy one year prior to trial treatment.
4. Presence of a chronic debilitating intestinal disease (e.g. Malabsorption, colonic tumor)

   a. Use of probiotics during FMT. Probiotics must be discontinued a minimum of 24 hours before FMT administration and patients are not permitted to take probiotics during the course of immunotherapy treatment.
5. Use of antibiotics within 2 weeks of enrollment in the study.
6. Presence of absolute contra-indications to FMT administration

   1. Toxic megacolon
   2. Severe dietary allergies (e.g. shellfish, nuts, seafood)
   3. Active inflammatory bowel disease
7. Expected to require any other form of systemic or localized anti-neoplastic therapy while on study.
8. Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for two years.

   a. NOTE: This time requirement does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
9. Active untreated central nervous system (CNS) metastases and/or leptomeningeal involvement (leptomeningeal enhancement on MRI/CT imaging and/or positive CSF cytology).
10. Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.

    a. Patients with vitiligo, type I diabetes, resolved childhood asthma/atopy are exceptions to this exclusion criteria.
11. A history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Has serious concomitant illnesses, such as: impaired cardiovascular function of clinically significant cardiovascular disease (uncontrolled congestive heart failure requiring treatment (NYHA grade > 2), uncontrolled hypertension, acute myocardial cardiac ischemia or unstable angina < 6 months prior to study entry, and severe cardiac arrhythmia), active systemic infections, and active inflammatory bowel disorders.

    a. This includes HIV or AIDS-related illness, or active HBV and HCV.
13. Has an active infection requiring systemic therapy.
14. Patient has received a live vaccine within 4 weeks prior to the first dose of treatment

    a. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in the NSCLC cohort by RECIST criteria. | up to 2 years
  Objective Response Rate (ORR) as defined by the proportion of patients with NSCLC whose Best Overall Response (BOR) is either a complete response (CR) or partial response (PR) as assessed by iRECIST, based on RECIST v1.1. BOR is defined as the best response designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy. CR or PR determinations included in the BOR assessment must be confirmed by a second scan performed no less than 4 weeks after the criteria for response are first met.

SECONDARY OUTCOMES:
Progression-free survival at 1 year in the NSCLC cohort by RECIST criteria. | At 3 and 6 months, then at 12 months and up to 2 years
  Progression-free survival (PFS) at 1 year as assessed by iRECIST and RECIST. PFS is defined by the proportion of treated subjects remaining progression-free and surviving at 1 year, defined as the time from registration to disease progression or death from any cause. The proportion will be calculated by the Kaplan-Meier estimate, which takes into account censored data.
Overall survival at 1 year in the NSCLC cohort assessed by RECIST criteria. | At 3 and 6 months, then at 12 months and up to 2 years
  Overall survival (OS) at 1 year as assessed by iRECIST and RECIST radiology, defined by OS will be defined as the time of patient registration to the time of death from any cause. The proportion will be calculated by the Kaplan-Meier estimate, which takes into account censored data.
Incidence of treatment-related adverse events (Safety and tolerability) | Safety follow-up will be maintained up to 90 days following the administration of the last study-drug dose.
  Safety of administration of FMT in combination with ICI in the Safety Analysis Dataset. The assessment of safety will be based on the incidence of AEs, SAEs, AEs leading to discontinuation, and deaths in the Safety Analysis dataset.
  Treatment-related adverse events will be graded according to the NCI CTCAE v5.0.
Incidence of treatment-related laboratory test abdnomarlities (Safety and tolerability) | Safety follow-up will be maintained up to 90 days following the administration of the last study-drug dose.
  Clinical laboratory test abnormalities will be examined. Laboratory values will be graded according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Elkrief, MD, Principal Investigator — CHUM
Locations (6):
- Canada (6):
  - London Health Sciences Centre, London, Ontario
  - DRCC Lakeridge Health, Oshawa, Ontario
  - Sunnybrook Health Sciences Centre/Sunnybrook Research Institute, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Québec, Centre intégré en cancérologie (CIC), Hôpital de L'Enfant-Jésus, Québec, Quebec

REFERENCES:
- [Derived] Duttagupta S, Messaoudene M, Hunter S, Desilets A, Jamal R, Mihalcioiu C, Belkaid W, Marcoux N, Fidelle M, Suissa D, Ponce M, Geiger M, Malo J, Piccinno G, Puncochar M, Filin A, Heidrich V, Rusu D, Mbaye B, Durand S, Ben Aissa I, Puller V, de Lahondes R, Blais N, Tehfe M, Owen S, Belanger K, Parvathy SN, Shieh B, Raphael J, Lenehan J, Breadner D, Rothenstein J, Rozza N, Maillou J, Nili S, Prifti DK, Pinto F, Armanini F, Kim-Schulze S, Marron TU, Kroemer G, Derosa L, Zitvogel L, Silverman M, Segata N, Vareki SM, Routy B, Elkrief A. Fecal microbiota transplantation plus immunotherapy in non-small cell lung cancer and melanoma: the phase 2 FMT-LUMINate trial. Nat Med. 2026 Jan 28. doi: 10.1038/s41591-025-04186-5. Online ahead of print. PMID 41606121